CLINICAL TRIAL: NCT05250648
Title: Phase IV Multicentric Clinical Trial to Evaluate the Efficacy of Hyperthermic Intraperitoneal Chemotherapy (HIPEC) with Mytomicin-C After Complete Surgical Cytoreduction in Patients with Colon Cancer Peritoneal Metastases
Brief Title: Clinical Trial on HIPEC with Mitomycin C in Colon Cancer Peritoneal Metastases (GECOP-MMC)
Acronym: GECOP-MMC
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitario de Fuenlabrada (Other)
Collaborators: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Principal Investigator, Fernando Pereira, Principal Investigator, Head of Surgery Dpt, Clinical Professor, Hospital Universitario de Fuenlabrada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GECOP-MMC; 2019-004679-37 (EudraCT Number)
Record Dates: First submitted 2022-01-23; First posted 2022-02-22 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Peritoneal Carcinomatosis; Colon Cancer
Keywords: HIPEC; Mitomycin; Colon Neoplasms; Peritoneal metastasis
MeSH Terms: conditions — Peritoneal Neoplasms; Colonic Neoplasms | interventions — Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Intervention Model Description: Recruitment will be carried out at the outpatient clinic, once the indication of CRS ± HIPEC (CC-PM of apparently limited volume without metastasis at other sites) has been established after presenting the case in the Multidisciplinary Tumour Board. Eligible patients need to meet the presurgical inclusion criteria (even though some criteria have to be confirmed during surgery for randomization), and sign the informed consent.
  Randomization occurs intraoperatively, once the extension of peritoneal disease is found to be truly limited (PCI ≤ 20) after complete surgical exploration, and only after radical surgery (CCS 0) has been possible. At this time, patients are randomized to receive HIPEC with MMC for 90 minutes (Arm 1), or no HIPEC and therefore surgery is finished (Arm 2).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- complete cytoreductive surgery plus HIPEC with Mytomicin C for 90 minutes (Active Comparator)
  Interventions: Drug: complete cytoreductive surgery plus HIPEC with Mytomicin C for 90 minutes
- complete cytoreductive surgery without HIPEC (Experimental)
  Interventions: Procedure: complete cytoreductive surgery without HIPEC

INTERVENTIONS:
Drug: complete cytoreductive surgery plus HIPEC with Mytomicin C for 90 minutes — In the arm with HIPEC, this will be performed with Mytomicin C, at a dose of 35 mg/m2 in peritoneal dialysis solution (2 liter/m2) for 90 minutes, with dose fractionation: 50% min 0, 25% min 30, 25% min 60
  Arms: complete cytoreductive surgery plus HIPEC with Mytomicin C for 90 minutes
Procedure: complete cytoreductive surgery without HIPEC — in the arm without HIPEC, only complete cytoreductive surgery will be performed
  Arms: complete cytoreductive surgery without HIPEC

SUMMARY:
The aim of this study is to assess whether there are differences in PERITONEAL RECURRENCE in patients with Colon Cancer Peritoneal Metastases treated with complete surgical resection and systemic chemotherapy, with (Group 1) or without (Group 2) HIPEC with Mitomycin-C.

DETAILED DESCRIPTION:
CytoReductive Surgery (CRS) + Hyperthermic IntraPEritoneal Chemotherapy (HIPEC), especially from the year 2000 onwards, has obtained unprecedented results in patients with low to moderate volume peritoneal metastases (PM) of colorectal cancer (CRC), so that it has gradually been accepted, even being considered the best treatment for these patients. However, the actual role of HIPEC as a necessary component of treatment is unknown, despite its proven experimental basis. The French PRODIGE 7 study, presented at ASCO in 2018 and published on January 2021, has raised doubts about the survival benefit of HIPEC. In this study, there was no difference in overall survival (OS) with or without HIPEC (with Oxaliplatin 30 minutes) after resection of PM-CRC. However, since its presentation, several methodological flaws have been identified: a short exposure time to Oxaliplatin, an overestimation of the effect of HIPEC on OS (18 months) considered for the sample calculation, or the choice of OS as the main endpoint (since HIPEC can reduce peritoneal relapses, while OS is also influenced by the systemic treatment received by all patients). Due to these shortcomings and some others, the results have not been assumed to be definitive. Therefore, the majority of units specialized in peritoneal surface malignancy, continue to consider HIPEC in these patients as a recommended option, usually changing Oxaliplatin for Mitomycin-C (MMC). With these premises we propose this multicenter Clinical Trial, correcting the retrospective defects of PRODIGE 7. To do this, the cytostatic used in HIPEC will be changed (MMC instead of oxaliplatin), the infusion time will be increased (from 30 to 90 minutes), rectal cancers are ruled out (only colon cancers will be included), cases with high peritoneal extension (PCI> 20) will be avoided, those cases in which a complete CRS (CCS 0) is not achieved will be excluded, and the main objective will be the Peritoneal Recurrence Free Survival (RFS) instead of the OS.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed colon adenocarcinoma, except signet ring cell carcinomas (those with > 50% of the tumor composed of these cells, which comprise only 1% of all colon adenocarcinomas).
2. Absence of previously treated or current extraperitoneal metastases, including distant lymphadenopathy (retroperitoneal, mediastinal, etc), liver metastases, or lung metastases (ruled out by PET-scan in case of doubt).
3. Synchronous or metachronous peritoneal metastasis of mild to moderate volume, with a PCI ≤ 20 (Appendix 2) (intraoperative confirmation).
4. Macroscopically complete surgical cytoreduction CCS-0 (intraoperative confirmation).
5. Treatment with perioperative systemic chemotherapy (SCT), before and/or after surgical procedure.
6. Age> 18 years.
7. Acceptable anesthetic/surgical risk: ASA 1-3 (Appendix 3), ECOG 0-1 (Appendix 4). No severe alterations in hematological, renal, cardiac, pulmonary or hepatic function (operable patients).
8. Information to the patient and signing of a study-specific informed consent.

Exclusion Criteria:

1. Peritoneal carcinomatosis of any other origin, particularly rectal cancer or appendicular adenocarcinoma, or signet ring cell colon cancer on histology.
2. No intraoperative confirmation of peritoneal disease (PCI 0). Likewise, cases of perianastomotic (local) or lymph node (locoregional) recurrences will be excluded.
3. High volume peritoneal disease with a PCI> 20 (intraoperative evaluation).
4. Concurrent or previously treated extraperitoneal disease.
5. Disease progression during preoperative chemotherapy, if received.
6. Patients previously treated with HIPEC.
7. History of other cancers (except cutaneous basal cell carcinoma or cervix carcinoma in situ) in the 5 years prior to entry into the study.
8. Patients included in another first-line clinical trial for the studied disease.
9. Pregnancy (or suspicion of it) or lactation period.
10. Emergency surgical intervention for obstruction or perforation of a primary tumour with synchronous PM (although rescue and secondary CRS + HIPEC after emergency surgery of the primary tumour are acceptable if inclusion criteria are fulfilled).
11. Persons deprived of liberty or under legal or administrative supervision.
12. Inability to understand the nature of the intervention, the risks, benefits, expected evolution and the need to undergo periodic medical examinations, either for geographical, social or psychological reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2022-03-02 (Actual); Primary Completion 2029-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Peritoneal Recurrence Free Survival | 3 years
  From the date of surgery to the date of peritoneal recurrence or death, or to the end of follow-up

SECONDARY OUTCOMES:
Global recurrence at any location (Disease Free Survival) | 3 years
  From the date of surgery to the date of recurrence at any site or death
Locoregional and distant recurrence rate (isolated or coincident, with or without simultaneous peritoneal recurrence) | 3 years
  From the date of surgery to the date of locoregional and/or distant recurrence
Postoperative complications (rate and severity grade) | days 1-90 after surgery
  Using the CTCAE v5.0 adverse event classification system, including those related to HIPEC.
Peritoneal and global recurrence rate according to stratified PCI | 3 years
  Rate of peritoneal and global recurrence in 3 subgroups of PCI ((1-10, 11-15, 16-20)
Overall survival | 3 years
  Months from from the day of treatment initiation (either neoadjuvant SCT or upfront CRS) to the date of death or to the end of follow-up.
Quality of Life with EORTC validated questionnaire Core 30 (QLQ-C30) | pre-surgery, at the end of postoperative SCT (an average 4-6 months), at 12 months and at 24 months
  The QLQ-CR29 is a supplementary questionnaire module to be employed in conjunction with the QLQ-C30. In fact, their numbering is consecutive (the last item of QLQ-C30 is number 30, being the first item of QLQ-CR29 number 31). Both have function and symptom scales/single-items. All of the scales and single-item measures range in score from 0 to 100. A high score for the functional scale and functional single-items represents a high level of functioning, whereas a high score for the symptom scales and symptom single-items represents a high level of symptomatology or problems.
Quality of Life with EORTC validated questionnaire Colorectal Cancer Module (QLQ-CR29). | pre-surgery, at the end of postoperative SCT (an average 4-6 months), at 12 months and at 24 months
  The QLQ-CR29 is a supplementary questionnaire module to be employed in conjunction with the QLQ-C30. In fact, their numbering is consecutive (the last item of QLQ-C30 is number 30, being the first item of QLQ-CR29 number 31). Both have function and symptom scales/single-items. All of the scales and single-item measures range in score from 0 to 100. A high score for the functional scale and functional single-items represents a high level of functioning, whereas a high score for the symptom scales and symptom single-items represents a high level of symptomatology or problems.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Pereira, PhD, Principal Investigator — Hospital Universitario de Fuenlabrada, Madrid, Spain
Locations (31):
- Spain (31):
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital Universitario Torrecárdenas, Almería, Almería
  - Complejo Hospitalario Universitario de Badajoz, Badajoz, Badajoz
  - Hospital Sant Joan Despi Moises Broggi, Sant Joan Despí, Barcelona
  - Hospital General Universitario de Castellón, Castellon, Castellón
  - Consorcio Hospitalario Provincial de Castellón, Castellon, Castellón
  - Hospital General Universitario de Ciudad Real, Ciudad Real, Ciudad Real
  - Hospital Universitario Reina Sofía, Córdoba, Córdoba
  - Hospital Universitario Donostia, San Sebastián, Gipuzkoa
  - Hospital Universitario de Gran Canaria Doctor Negrín, Las Palmas de Gran Canaria, Gran Canaria
  - Hospital Universitario Principe de Asturias, Alcalá de Henares, Madrid
  - Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid
  - HOSPITAL UNIVERSITARIO DE FUENLABRADA (Coordinating Centre), Fuenlabrada, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid, Madrid
  - Md Anderson Cancer Center, Madrid, Madrid
  - Hospital Universitario Ramón Y Cajal, Madrid, Madrid
  - Fundación Jiménez Díaz, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital Universitario Infanta Elena, Valdemoro, Madrid
  - Hospital Universitario Son Espases, Palma de Mallorca, Mallorca
  - Hospital Universitario Virgen de La Arrixaca, El Palmar, Murcia
  - Hospital General Universitario Reina Sofía, Murcia, Murcia
  - Hospital Quirónsalud Málaga, Málaga, Málaga
  - Hospital Regional Universitario de Málaga, Málaga, MÁLAGA
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario Virgen Del Rocío, Seville, Sevilla
  - Instituto Valenciano de Oncología, Valencia, Valencia
  - Hospital Clinico Universitario de Valencia, Valencia, Valencia
  - Hospital Universitario Y Politécnico La Fe, Valencia, Valencia
  - Hospital Universitario Río Hortega, Valladolid, Valladolid
  - Hospital Clínico Universitario "Lozano Blesa", Zaragoza, Zaragoza

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication, after deidentification (text, tables, figures and appendices) With whom? Researchers who provide a methodologically sound proposal. For what types of analyses? for individual participant data meta-analysis.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will be available beginning 9 months and ending 36 months following article publication
Access Criteria: To obtain the data, a proposal must be sent to fernando.pereira@salud.madrid.org. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Background] Pereira F, Serrano A, Manzanedo I, Perez-Viejo E, Gonzalez-Moreno S, Gonzalez-Bayon L, Arjona-Sanchez A, Torres J, Ramos I, Barrios ME, Cascales P, Morales R, Boldo E, Garcia-Fadrique A, Arteaga X, Gutierrez-Calvo A, Sanchez-Garcia S, Asensio E, Ramirez CP, Artiles M, Vaque J, Parra PA, Villarejo P, Munoz-Casares C, Turienzo E, Calero A, Torrejimeno IJ, Prieto I, Galindo J, Borrego V, Marcello ME, Rihuete C, Carrasco J, Gomez-Quiles L. GECOP-MMC: phase IV randomized clinical trial to evaluate the efficacy of hyperthermic intraperitoneal chemotherapy (HIPEC) with mytomicin-C after complete surgical cytoreduction in patients with colon cancer peritoneal metastases. BMC Cancer. 2022 May 12;22(1):536. doi: 10.1186/s12885-022-09572-7. PMID 35549912